CLINICAL TRIAL: NCT00183690
Title: Treating Terror-Related PTSD in Adolescents
Brief Title: Prolonged Exposure Therapy Versus Active Psychotherapy in Treating Post-Traumatic Stress Disorder in Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Eva Gilboa-Schechtman, Bar-ILan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH071660 (NIH); DATR AD-TS
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2008-12-12 (Estimated); Status verified 2008-12

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD; Anxiety Disorder; Trauma; Adolescents; Cognitive Behavioral Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants receiving prolonged exposure therapy
  Interventions: Procedure: Prolonged Exposure Therapy
- 2 (Active Comparator): Participants receiving active psychotherapy
  Interventions: Procedure: Active Psychotherapy

INTERVENTIONS:
Procedure: Prolonged Exposure Therapy — Prolonged exposure therapy includes a trauma focused protocol and cognitive behavioral treatment for PTSD. Cognitive behavioral treatment includes psychoeducation, in vivo exposures, and imaginal exposures.
  Arms: 1
Procedure: Active Psychotherapy — Active psychotherapy includes non-trauma focused therapy, based on time-limited psychodynamic treatment, which includes a formulation of a central issue and open-associative sessions exploring main conflicts and drives.
  Arms: 2

SUMMARY:
This study will compare the effectiveness of prolonged exposure therapy versus active psychotherapy in treating post-traumatic stress disorder (PTSD) in adolescents.

DETAILED DESCRIPTION:
PTSD is an anxiety disorder that can develop after exposure to an event in harm to the life or physical integrity of oneself or others has occurred or was threatened. People with PTSD have persistent frightening thoughts and memories of their ordeal and often feel emotionally numb, especially with people to whom they were once close. Effective treatments for post-traumatic stress disorder are available, and research is yielding new, improved therapies that can help reduce symptoms of PTSD. Prolonged exposure (PE) therapy is a brief cognitive behavioral therapy that has been effective in treating symptoms of PTSD in adults. However, no treatments have been proven effective for the treatment of PTSD in adolescents. This study will compare the effectiveness of PE therapy versus non-trauma directed active psychotherapy in reducing the symptoms of PTSD in adolescents. In addition, this study aims to refine the existing PE treatment protocol for adolescents with PTSD.

Participants in this single-blind study will be randomly assigned to receive either PE therapy or AP. All participants will receive 12 to 18 therapy sessions, which will be conducted weekly. Assessments of PTSD symptoms, depression, and overall functioning will be conducted at baseline, immediately post-treatment, and 3 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of PTSD
* In grades 6-12
* No change in medication regimen for more than 6 weeks

Exclusion Criteria:

* Diagnosis of ADHD, conduct disorder, thought disorder, or bipolar disorder

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2004-09; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Symptoms of post-traumatic stress disorder | Measured at Month 3
Symptoms of depression | Measured at Month 3

SECONDARY OUTCOMES:
Clinical global assessment of overall functioning | Measured at Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Eva Gilboa-Schechtman, PhD, Principal Investigator — Bar Ilan University; Edna B. Foa, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Schneider Children's Medical Center of Israel, Petach Tikvah, Israel

REFERENCES:
- [Derived] Gilboa-Schechtman E, Foa EB, Shafran N, Aderka IM, Powers MB, Rachamim L, Rosenbach L, Yadin E, Apter A. Prolonged exposure versus dynamic therapy for adolescent PTSD: a pilot randomized controlled trial. J Am Acad Child Adolesc Psychiatry. 2010 Oct;49(10):1034-42. doi: 10.1016/j.jaac.2010.07.014. Epub 2010 Sep 6. PMID 20855048